CLINICAL TRIAL: NCT02607995
Title: Structured Psychoeducation for Unemployed Adolescents With Extreme Obesity in a Multicenter Observational Study Focusing on Feasibility
Acronym: STEREOplus
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: Center for Sepsis Control and Care, Germany (Other); Zentrum für klinische Studien Essen (Other); JobCenter Essen Mitte (Other); Jobcenter Bottrop (Other); Jobcenter Gelsenkirchen (Other); Jobcenter Oberhausen (Other); Jobcenter Mülheim an der Ruhr (Other); Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Martin Wabitsch, Prof. Dr., University of Ulm
Other Study IDs: U1111-1131-4384f
Record Dates: First submitted 2015-09-28; First posted 2015-11-18 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Extreme Obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- low key intervention: for the whole group
  Interventions: Behavioral: Behavioral standardized manual-based multidisciplinary routine care

INTERVENTIONS:
Behavioral: Behavioral standardized manual-based multidisciplinary routine care — Behavioral standardized manual-based multidisciplinary routine care (lifestyle intervention). Six sessions offered over the course of three to six months with a focus on weight loss. The topics 1) causes, consequences and treatment options of obesity, 2) nutrition, 3) eating behaviors and problem solving strategies, 4) self esteem and emotional eating, 5) exercise, and 6) use of media will be covered.

SUMMARY:
Obesity occurs more frequently in subjects of a lower socioeconomic status and is associated with a lower income and unemployment. On the other hand, there is limited access of individuals with low socioeconomic status to conventional obesity treatments and bariatric surgery.

In STEREOplus the investigators will ascertain unemployed adolescents with obesity and extreme obesity at five job centers in the Ruhr area. Unemployed obese youths and young adults (BMI ≥ 30kg/m2) between the ages of 14 and 24.9 years are eligible to participate. Participants will be asked to complete a series of questionnaires on their general health, psychosocial situation and wellbeing, and will be offered a thorough medical evaluation. Individuals who complete the baseline evaluations will be invited to participate in six group sessions of conventional obesity treatment over a three months period. After six months, participants will complete further questionnaires to evaluate the effects of the interventions on quality of life and psychosocial functioning. Weight status (BMI) will also be measured. Adolescents who attended at least five sessions and are interested in bariatric surgery will have access to a structured information and preparation program for bariatric surgery.

The overall objective of STEREOplus is to generate data on the feasibility of the planned implementation of a treatment targeted to a high risk group with a low socioeconomic background in order to reduce treatment barriers.

DETAILED DESCRIPTION:
Obesity occurs more frequently in subjects of a lower socio-economic status and is associated with a lower income and unemployment. Besides the obesity-related impairments in daily life, stigmatisation additionally aggravates the difficulties of vocational integration by multiple disadvantages in the process of application for employment, job interviews and performance evaluation. On the other hand, there is limited access of individuals with low socioeconomic status to conventional obesity treatments and bariatric surgery.

In this multicenter observational study, the investigators aim to assess the acceptance of a manual based low key group intervention targeted at unemployed adolescents (BMI≥30 kg/m2; 14-24 years old) recruited on the premises of five local job centers in the Ruhr area. The study is part of the "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care", short: "Youth with extreme obesity Study (YES), which also comprises the recruitment and characterization of obese (BMI 30-34.9kg/m2) and extremely obese (BMI ≥ 35kg/m2) youth from different healthcare- and non healthcare settings, a structured prospective evaluation of adolescent bariatric surgery, economic assessments of the financial burden of extreme adolescent obesity on the healthcare system, and a long-term prospective observation study.

The participating job centers are located in five cities in the West (Ruhr-Area). The investigators will screen 300 unemployed adolescents aged 14 to 24.9 years with obesity and extreme obesity (BMI ≥30kg/m2) over a 24 month period. A total of 80 subjects will be enrolled. Baseline assessments include an array of standardized questionnaires and validated instruments to assess health, psycho-social situation, psychiatric co-morbidities and health related quality of life, as well as an in-depth medical evaluation.

Individuals who complete the baseline evaluations will be invited to participate in six group sessions over a three month period. Adolescents who attended at least five sessions and are interested in bariatric surgery will have access to a structured information and preparation program for bariatric surgery. The adherence and effects of the interventions on BMI, health related quality of life and psycho-social functioning will be assessed via questionnaires after six months. All statistical analyses will be exploratory/descriptive. The project will reveal the feasibility of the implementation of the described intervention approach focusing on reducing treatment barriers for unemployed adolescents with obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2
* written informed consent
* sufficient knowledge of the German language to participate in the intervention
* participation in subproject 1

Exclusion Criteria:

* any psychiatric disorder that requires inpatient treatment (e.g. psychotic disorder, severe depression with suicidal behavior)
* IQ < 70

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: obese adolescents or young adults presenting at 5 different job centers
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Change in BMI | baseline and 6 months
  The BMI will be measured and compared
Adherence measured as the participation rate in the intervention | 6 months
  Adherence will be measured as the participation rate in the intervention
Change in participation rate in the first and second labor market | baseline and 6 months
  The number of patients able to integrate themselves into the job market will be assessed

SECONDARY OUTCOMES:
Change in quality of life (DISABKIDS) | baseline and 6 months
  The 37 item DISABKIDS questionnaire will be applied twice, and the score difference in each of the 6 subscales will be calculated for each subject
Change in depression score (Beck Depression Inventory-II) | baseline and 6 months
  The Becks Depression Inventory 2 questionnaire will be applied twice, and the score difference will be calculated for each subject. Answers will be reviewed immediately to identify and treat subjects at risk for self harm
Change in self-esteem (Rosenberg scale) | baseline and 6 months
  The Rosenberg´s scale patient questionnaire will be applied twice, and the score difference will be calculated for each subject
Change in perceived stress (PSQ Fliege scale) | baseline and 6 months
  The Fliege scale questionnaire will be applied twice, and the score difference will be calculated for each subject
Change in somatic and psychiatric disorders (standardized patient questionnaire) | baseline and 6 months
  The occurrence of somatic and psychiatric disorders will be assessed twice via a standardized patient questionnaire, and changes evaluated for each patient
Change in self-reported physician and therapist contact (standardized patient questionnaire) | baseline and 6 months
  The frequency of self-reported physician and therapist contact will be elicited twice via standardized patient questionnaire (modified after KIGGS and TeenLABS) and the difference will be calculated for each subject
Change in self-reported time spent outside the home (standardized patient questionnaire) | baseline and 6 months
  The self-reported time spent outside the home will be elicited twice via standardized patient questionnaire (modified after KIGGS and TeenLABS) and the difference will be calculated for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Hebebrand, Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen
Locations (1):
- University Duisburg-Essen, Essen, Germany